CLINICAL TRIAL: NCT04442815
Title: Analysis of Patient Ventilator Asynchrony Using Electrical Impedance Tomography (EIT) in Patients With Acute Respiratory Failure
Brief Title: EIT in Patient Ventilator Asynchrony
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Wen Chen, Associate professor and attending physician, National Cheng-Kung University Hospital
Other Study IDs: EIT and ARF
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: ARDS, Human
Keywords: ARDS, patient-ventilator interaction, EIT
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Patient-ventilator asynchrony is an important clinical issue in mechanically ventilated patients. For patients with moderate to severe acute respiratory distress syndrome (ARDS), various types of patient ventilator asynchrony may lead to injury of the lung. For example, double cycling may lead to high tidal volume and pendelluft may result in transient overstretch of dependent lung region. In this project, the investigators will record and analyze various types of patient-ventilator asynchrony in ARDS patients and analyze the regional distribution of lung gas and determined their harmful effect via concomitant recording of EIT and transpulmonary pressure. The results may influence our ventilator management of ARDS patients.

DETAILED DESCRIPTION:
Patients and Methods:

Admitted ventilated patients who are greater than 18 years old and fulfilled the Berlin's diagnostic criteria of moderate to severe ARDS will be selected to enter our study. The exclusion criteria include (1) patients with metallic materials in the body (including wire, pin or implanted electrical devices etc.); (2) patients with cutaneous diseases which prohibited the application of electrode leads to attached the body; (3) severe chronic obstructive pulmonary diseases; (4) hemodynamically unstable; (5) proved barotrauma (including pneumothorax or pneumomediastinum etc.); (6) pregnancy; (7) diseases characterized with increased intracranial pressure; (8) patients or family who refused the informed consent. All patients who fulfilled the diagnosis of ARDS will receive standard care of low tidal volume ventilator therapy. The tidal volume 6 ml/Kg will be used. The investigators expect to enroll at least 20 analyzable cases. Sedation and paralysis are usually used in moderate to severe ARDS patients and daily interruption of sedation and paralysis is a standard practice. The investigators will perform recording during daily interruption of sedation and paralysis, up to 60 minutes period will be recorded during the interruption period. Recording will be done at least once for registered case and could be repeated in case of unsatisfactory signals.

Instrumentation In all patients, air flow will be measured using a pneumotachograph (Hamilton AG, or Hans Rudolf) connected to a differential pressure transducer (MP 45, Validyne Corp., Northridge, CA). The flow sensor will be placed between the endotracheal tube and the Y-piece of the ventilator. Tidal volume will be obtained by integrating the flow signal. Airway pressure and esophageal pressure will be measured using differential pressure transducers (P300D, Validyne Corp., Northridge, CA.). An appropriate esophageal pressure signal will be confirmed according to the standard guideline[27]. All signals are sampled and digitalized at 200 Hz and data are stored in a data acquisition system (MP150, Acqknowledgement, Biopac, Goleta, CA).

Measurements:

Electrical impedance tomography:

The investigators use a commercial EIT monitor (PulmoVista 500, Drager Medical GmbH, Lubeck, Germany). An electrode belt with 16 equally spaced electrodes will be placed around the patient's thorax at the 4th to 5th intercostal space. Impedance data will be acquired by applying adjacent alternate current injection (50 KHz) and measuring the voltage difference between the adjacent leads and a finite element method-based, linearized Newton-Raphson reconstruction algorithm is used to construct the impedance data. The PulmoVista 500 monitor displays functional EIT images, i.e. relative impedance changes including tidal ventilation and end-expiratory lung impedance (EELI) changes. During the study phases, EIT data will be registered at 20-40 Hz and low-pass filtered (35 per minute) and stored for offline analysis.

The individual impedance recording (10 minutes per segment) will be linked into a single file and impedance calculation will thus be done off-line. The investigators will subdivide the impedance recordings into ventral to dorsal parts. The investigators define the presence of pendelluft as the presence of opposite impedance change (△Z) between dependent and independent zones during a breathing effort. The breath could occur in inspiration phase, expiratory phase or in transition. Estimation of volume of pendelluft will be determined by the integrated volume and corresponding impedance change.

Respiratory mechanics:

The investigators will record the peak and plateau airway pressure, total PEEP, flow and the esophageal pressure. Transpulmonary pressure (PL) will be calculated as the difference between Paw and Pes calculate the transpulmonary pressure.

Study protocol The investigators target at moderate to severe ARDS patients who are already under deep sedation with neuromuscular blockade. As daily interruption of sedatives and muscle relaxant are routinely performed in our ICU, we will record the respiratory mechanics and EIT data for about one hour which should include both controlled and spontaneous breathing period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe ARDS

Exclusion Criteria:

* Severe chronic obstructive pulmonary diseases
* Proved barotrauma (including pneumothorax or pneumomediastinum etc.);
* Pregnancy
* Diseases characterized with increased intracranial pressure
* Patients or family who refused the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all genders except pregnant woman
Study Population: moderate to severe ARDS patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Patient ventilator asynchrony | up to 1 hour following interruption of muscle relaxant
  Various types of patient ventilator asynchrony
Regional ventilation distribution by EIT | up to 1 hour following interruption of muscle relaxant
  Regional ventilation distribution by EIT in various types of patient ventilator asynchrony

SECONDARY OUTCOMES:
hospitalization day and final outcome | up to 3 months
  duration of hospitalization and hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Wen Chen, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Chang-Wen Chen, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared once the data is published